CLINICAL TRIAL: NCT06880354
Title: A Clinical Study to Evaluate the Safety and Efficacy of CLL1 and CD38 Dual-Target CAR-T Cell Injection in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024059
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention（CLL1 and CD38 Dual-Target CAR-T Cell Injection） (Experimental): This study is a single-center open-label clinical study. The main purpose is an IIT clinical trial to evaluate the safety and preliminary efficacy of CLL1 and CD38 dual CAR-T injection in r/r AML subjects . The enrolled subjects were patients with relapsed and refractory acute myeloid leukemia (r/r AML) .
  Interventions: Drug: CLL1 and CD38 Dual-Target CAR-T Cell Injection

INTERVENTIONS:
Drug: CLL1 and CD38 Dual-Target CAR-T Cell Injection — This product is a lentiviral gene-modified autologous chimeric antigen receptor T-cell product that targets both CLL1 and CD38.

SUMMARY:
This is a single-arm, open-label, phase I dose-escalation clinical study to evaluate the safety and preliminary efficacy of CLL1 and CD38 dual-target CAR T cell injection in r/r AML subjects.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase I dose-escalation clinical study to evaluate the safety and preliminary efficacy of CLL1 and CD38 dual-target CAR T cell injection in r/r AML subjects.

The main purpose of this study is to evaluate the safety of CLL1 and CD38 dual - target CAR - T cell injection in the treatment of r/r AML and the study contains two phases with the first phase adopting an ATD design and the second phase adopting a 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent, 18-70 years old (including the critical value);
2. Diagnosed with acute myeloid leukemia (except for APL) based on the World Health Organization (WHO) 2022 criteria and meeting the diagnostic criteria for relapsed/refractory AML (refer to the 2023 Chinese Guidelines for the Diagnosis and Treatment of relapsed refractory acute myeloid leukemia);
3. Positive expression of CLL1 and/or CD38 in tumor cells;
4. Estimated survival ≥3 months;
5. Have a confirmed donor for allogeneic hematopoietic stem cell transplantation. After the CAR-T cells were infused, subjects could undergo potential allogeneic hematopoietic stem cell transplantation at any time;
6. ECOG score of 0~2 during the screening phase;
7. Adequate functional reserve of organs:

   1. Alanine aminotransferase/aspartate aminotransferase ≤2.5× ULN;
   2. Total serum bilirubin ≤2× ULN, except in subjects with congenital bilirubinemia (direct bilirubin ≤1.5× ULN in subjects with Gilbert's syndrome);
   3. Serum creatinine clearance > 45mL/min (calculated according to Cockcroft-Gault formula);
   4. Left ventricular ejection fraction (LVEF) ≥45%;
   5. Basal finger oxygen saturation ≥92% in room air.
8. The ability to discontinue corticosteroids (dexamethasone ≥3mg/ day or other equivalent dose of hormones) from day 7 and continue until 30 days after CAR T cell infusion;
9. Pregnant women of childbearing potential should be negative for HCG (immunofluorescence) tests during screening and baseline. Male subjects must agree not to donate sperm for at least two years after the infusion. Male subjects and his sexual partner with childbearing potential must agree to use highly effective contraception for at least 2 years after the infusion;
10. Agree to follow-up in accordance with the protocol and the requirements outlined in the informed consent form;
11. Voluntarily sign the ICF.

Exclusion Criteria:

1. Known allergy to any of the drug ingredients to be used in this study;
2. With a history of the following concomitant treatments:

   1. Received a cumulative dose of prednisone (or equivalent corticosteroids). Greater than or equal to ≥ 70 mg within 7 days prior to apheresis;
   2. Based on the investigator's assessment, there is a comorbidity that requires the use of systemic corticosteroids (≥ 70 mg total dose of prednisone or equivalent doses of other corticosteroids) or other immunosuppressive medications within 12 weeks after the study treatment;
   3. Received systemic anti-tumor therapy within 14 days before apheresis or within five half-lives of the drug, whichever was shorter, including but not limited to cytotoxic therapy, targeted therapy, or an investigational drug treatment;
   4. Received radiotherapy 4 weeks before apheresis;
   5. Received donor lymphocyte infusion within 6 weeks before apheresis.
3. Acute promyelocytic leukemia was diagnosed;
4. Have previously been received CAR-T therapy, CAR-NK therapy or any other genetically modified cell therapy;
5. Received allogeneic hematopoietic stem cell transplantation within 6 months before screening phase;
6. Active graft-versus-host disease (GvHD) at the time of screening or active acute or chronic GvHD within 4 weeks of enrollment or the need for immunosuppressive drugs;
7. An active infection that requires systemic treatment;
8. Any history of active malignancy (excluding non-melanoma skin cancer, cervical carcinoma in situ, bladder cancer, breast cancer, or other similar cancers, with a disease-free survival period of more than 5 years and no signs of recurrence after curative treatment);
9. Experienced a stroke or seizure within 6 months prior to signing the ICF;
10. Presence of any heart diseases as follows:

    1. New York Heart Association (NYHA) Stage III or IV heart failure;
    2. Myocardial infarction or coronary artery bypass graft (CABG) ≤ 6 months prior to enrollment;
    3. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree II-III atrioventricular block, and electrocardiographic corrected QTcF interval ≥480 ms;
    4. History of severe non-ischemic cardiomyopathy;
    5. Cardiac dysfunction (LV <45%), as assessed by echocardiography or multigated acquisition scanning, or other clinically symptomatic cardiac disease within 6 months before enrollment;
    6. Clinically uncontrolled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100mmHg) (based on the mean of ≥2 measurements).
11. Active or past central nervous system involvement, or clinical manifestations of central involvement in acute myeloid leukemia;
12. Any positive results of the following virological test results:

    1. Human immunodeficiency virus antibodies (HIV antibodies);
    2. Hepatitis B surface antigen (HBsAg) positive; Or hepatitis B core antibody (HBcAb) positive, and hepatitis B virus (HBV) -DNA copy number higher than the lower limit of detection;
    3. Hepatitis C virus antibody positive, and hepatitis C virus RNA higher than the lower limit of detection;
    4. Treponema pallidum antibody (TPPA antibody).
13. There is pulmonary fibrosis;
14. With active autoimmune diseases (e.g. systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, etc.);
15. Received live attenuated vaccine within 4 weeks prior to screening;
16. Receipt of major surgery within 4 weeks prior to apheresis or a plan to receive surgeries during the study (except for diagnostic biopsy);
17. Pregnant women or nursing women who do not agree to give up breastfeeding, men and women who plan to have children during the study period or within 2 years after receiving the study treatment;
18. Acute side effects caused by previous treatment did not return to grade 1 or below (except those that the investigators judged to have no safety risk, such as hair loss, stable hypothyroidism after hormone replacement therapy, etc.);
19. According to the investigator's judgment, conditions that interfere with the subject's participation in the entire trial, confound the trial results, or make participation in the trial not in the best interest of the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) Rate | 28 days
  Proportion of subjects with DLT within 28 days after infusion of CLL1/CD38 dual-target CAR-T cell injection.
Adverse Events （AEs） | 96 weeks
  Proportion of subjects experiencing AE within 96 weeks after infusion of CLL1/CD38 dual-target CAR-T cell injection.

SECONDARY OUTCOMES:
Complete Remission Rate (CRc) | 96 weeks
  Proportion of subjects achieving CR + CR with partial hematologic recovery (CRh) +CR with incomplete hematologic recovery (CRi) (Patients achieving CRh are no longer repeatedly recorded as CRi).
Overall Response Rate (ORR) | 96 weeks
  Proportion of subjects achieving CR+CRi+CRh+MLFS+PR.
MRD negative rate and MRD negative duration | 96 weeks
  MRD negative proportion and MRD negative duration in CR/CRh/CRi subjects were measured by qPCR and/or flow cytometry.
Duration of Remission（DOR） | 96 weeks
  The time from CR/CRh/CRi first assessed to disease recurrence or death from any cause.
Event-free Survival (EFS) | 96 weeks
  The time from receiving CAR-T cell infusion to treatment failure, disease relapse, or death from any cause (whichever occurs first).
Overall Survival (OS) | 96 weeks
  The time from cell infusion to death from any cause was calculated.
Indicators of proliferation and survival in vivo | 96 weeks
  The number of CAR gene copies and CAR-T cells in bone marrow and peripheral blood after receiving CAR-T cell infusion.
Anti-drug Antibodies | 96 weeks
  Proportion of subjects who developed anti-drug antibodies in peripheral blood after CAR-T cell injection infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, China, Tianjin, China